CLINICAL TRIAL: NCT03516253
Title: Fish Oil and Evening Primrose Oil in the Treatment of Breast Cancer
Brief Title: Fish Oil and EPO in Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Aleksandra Arsic, Research Associate Professor, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: VMA-253-18
Record Dates: First submitted 2018-03-06; First posted 2018-05-04 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fish Oils

STUDY DESIGN:
Intervention Model Description: This study is a parallel, randomized, double blind, controlled, 3-months supplementation, investigating health effects of dietary intake of fish oil and EPO, in patients with breast cancer undergoing chemotherapy.
  At the beginning of the study, all patients received nutritional counseling, where half of the study subjects are randomly assigned to a treatment arm with fish oil and EPO, or control arm with mineral oil as placebo. Treatment arm is provided with 2 gel capsules of fish oil and 3 gel capsules of EPO (400 mg eicosapentaenoic acid, 600 mg docosahexaenoic acid and 351 mg gamma-linolenic acid). Control arm will consume 5 gel capsules of 1g of mineral oil.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Dietary Supplement: Fish oil + EPO. Fish oil (2 gel capsules, each 1g fish oil with 500 mg EPA+DHA) and EPO (Evening primrose oil 3 gel capsules with 117 mg GLA), 3 months with lunch.
  Interventions: Dietary Supplement: Fish oil + EPO
- Control group (No Intervention): Dietary Supplement: Mineral oil (5 gel capsules, each 1g mineral oil), 3 months with lunch.

INTERVENTIONS:
Dietary Supplement: Fish oil + EPO — Supplementation with both fish oil and EPO
  Arms: Intervention group

SUMMARY:
Recent literature data suggest beneficial effects of dietary fats in patients with cancers, in particular polyunsaturated fatty acids (PUFAs). Fish oil and evening primrose oil provide a high amount of PUFAs and a desirable n-6/n-3 PUFAs ratio.

DETAILED DESCRIPTION:
Breast cancer (BC) is leading cancer in women. As most of the cancers, it is characterized by inflammation and alternations in lipid and fatty acid metabolism. Patients with BC have impaired fatty acid profiles, low level of PUFAs, and high n-6/n-3 PUFAs ratio. Moreover, these changes are related to clinical outcome.

Fish oil is the richest source of anti-inflammatory n-3 PUFAs. Evening primrose oil (EPO) is rich in 18:3 n-6, the only n-6 fatty acid with an anti-inflammatory effect. Dietary intake of fish oil or EPO has been shown to decrease inflammation and improve PUFAs status in patients with cancers. However, it is not known what is the effect of combined EPO and fish oil in BC patients.

The study design is double-blind, controlled, randomized nutritional intervention. The participants are randomly assigned into intervention and control group before starting chemotherapy. All patients receive nutritional counseling to achieve a daily energy and protein intake according to recommended dietary allowances, with (intervention) or without (control) of milled seed mix.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer,
* Clinical Stadium III and IV,
* Patients able to understand requirements of the study and provide written informed consent-

Exclusion Criteria:

* Previous radio- or chemotherapy
* Other serious chronic diseases
* Statin therapy
* Use of fat-based dietary supplements (such as fish oil, evening primrose oil etc) 3 months prior to study

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-20 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Change in disease status | Baseline, 3 months, 1 year
  Remission, stable disease or progression
Change in quality of life | Baseline, 3 months, 1 year
  Assessed by standardized questionnaires, scale 1-4 (1-not at all, 2- a little, 3 - quite a bit, 4- very much), higher value represents worse outcome.

SECONDARY OUTCOMES:
Changes in nutritional status | Baseline, 3 months, 1 year
  Changes in body weight measured by bio-impedance analyzer, from baseline to endpoint
Changes in lipid profiles | Baseline, 3 months, 1 year
  Changes in lipid profiles (cholesterol, HDL, LDL and triglycerides) from baseline to endpoint
Changes in plasma fatty acids profiles | Baseline, 3 months, 1 year
  Changes in plasma fatty acids profiles from baseline to endpoint
Changes in interleukins | Baseline, 3 months, 1 year
  Changes in interleukins (IL)-6, 8,10 and TNF alpha from baseline to endpoint
Changes in activity of superoxide dismutase. | Baseline, 3 months, 1 year
  Measures of activity of superoxide dismutase.
Changes in activity of catalase. | Baseline, 3 months, 1 year
  Measures of activity of catalase.
Changes in activity of glutathion peroxidase. | Baseline, 3 months, 1 year
  Measures of activity of glutathion peroxidase.
Changes in activity of glutathion reductase. | Baseline, 3 months, 1 year
  Measures of activity of glutathion reductase.

CONTACTS AND LOCATIONS:
Locations (2):
- Serbia (2):
  - Military medical academy, Belgrade
  - University of Belgrade, Belgrade

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arsic A, Krstic P, Paunovic M, Nedovic J, Jakovljevic V, Vucic V. Anti-inflammatory effect of combining fish oil and evening primrose oil supplementation on breast cancer patients undergoing chemotherapy: a randomized placebo-controlled trial. Sci Rep. 2023 Apr 20;13(1):6449. doi: 10.1038/s41598-023-28411-8. PMID 37081029